CLINICAL TRIAL: NCT01624935
Title: Randomized Controlled Clinical Trial of Interpersonal Therapy for Survivors of the Sichuan Earthquake
Brief Title: Clinical Trial of Interpersonal Therapy for Survivors of the Sichuan Earthquake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10-02408
Record Dates: First submitted 2012-02-07; First posted 2012-06-21 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Posttraumatic Stress Disorder; Depression
Keywords: PTSD; earthquake; disaster; global mental health; disaster mental health; depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- psychotherapy (Experimental): psychotherapy
  Interventions: Behavioral: interpersonal psychotherapy
- treatment as usual (Other): TAU control
  Interventions: Behavioral: interpersonal psychotherapy

INTERVENTIONS:
Behavioral: interpersonal psychotherapy — interpersonal psychotherapy

SUMMARY:
The enormous global burden of mental illness has been estimated through the publication of the Global Burden of Disease Study. Research confirms that populations exposed to mass trauma such as natural disaster bear a particularly high burden of mental disorders, with depression and Posttraumatic Stress Disorder (PTSD) generally being the top two adult psychiatric diagnoses. In traumatized populations, these disorders do not remit with replacement of material losses or resettlement to safe locations, but rather tend to become chronic conditions with attendant disability. PTSD and depression are risk factors for anger, interpersonal discord and violence, not only among those who have trauma and depression, but also among their spouses and children. This "infectious" model of trauma/violence is critically important in the setting of natural disaster, as increased levels of interpersonal violence within the afflicted community hinder its recovery. To date, there has been little research on the interpersonal effects of mass trauma. The proposed research is a randomized controlled trial of "Interpersonal Therapy" (IPT) versus wait list control (WLC) for survivors of the Sichuan Earthquake living in Shifang, China. IPT, a very effective therapy for depression, has been adapted for PTSD treatment and developing country settings. Measures will evaluate success of the treatment not only in terms of individual depression and PTSD symptoms, but also with respect to interpersonal functioning.

Hypothesis 1: Relative to wait list control, fewer subjects who received IPT will meet criteria for Depression and PTSD at the conclusion of the RCT.

Hypothesis 2: Subjects who received IPT will have greater improvement of social functioning than wait list controls.

DETAILED DESCRIPTION:
Interpersonal Psychotherapy adapted for local mental health care needs was applied using wait list control design.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years;
* diagnosis with Depressive Disorder and Posttraumatic Stress Disorder (PTSD);
* Ability to attend weekly therapy sessions for 12 weeks and return for post-treatment screening;
* Ability to give verbal informed consent

Exclusion Criteria:

* Cognitive dysfunction which requires a higher level of care and/or interferes with ability to participate in IPT;
* Severe thought or mood disorder symptoms which requires a higher level of care and/or interferes with ability to participate in IPT;
* drug and alcohol dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | baseline through week 24
  CAPS and SCID assessed before and after treatment after tx conclusion at week 0, week 12, week 24

SECONDARY OUTCOMES:
Standard Clinical Interview for DSM IV Diagnosis (SCID) | baseline through week 24
  CAPS and SCID assessed before and after treatment after tx conclusion at week 0, week 12, week 24

CONTACTS AND LOCATIONS:
Overall Officials: Susan Meffert, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Wuhan Hospital for Psychotherapy, Fangting, Sichuan, China

REFERENCES:
- [Derived] Jiang RF, Tong HQ, Delucchi KL, Neylan TC, Shi Q, Meffert SM. Interpersonal psychotherapy versus treatment as usual for PTSD and depression among Sichuan earthquake survivors: a randomized clinical trial. Confl Health. 2014 Sep 4;8:14. doi: 10.1186/1752-1505-8-14. eCollection 2014. PMID 25254070